CLINICAL TRIAL: NCT06511921
Title: Early Versus Late Biologic Therapy for Post-operative Perforated Crohn's Disease Patients
Brief Title: Effect of Biologic Therapy on Surgical Outcomes for Perforated Crohn's Patients
Status: Completed | Type: Observational
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Reham Zakaria Mohamed Ahmed, lecturer of general surgery, Zagazig University
Other Study IDs: #479\9-July-2024
Record Dates: First submitted 2024-07-12; First posted 2024-07-22 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2024-07

CONDITIONS: Crohn Disease
Keywords: perforation; biologic therapy; ileostomy
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- post operative Crohn's patients
  Interventions: Biological: early biologic therapy
- post operative Cronn's patients
  Interventions: Biological: late biologic therapy

INTERVENTIONS:
Biological: early biologic therapy — biologic therapy for perforated Crohn's disease in the early postoperative period
  Groups: post operative Crohn's patients
Biological: late biologic therapy — no biologic therapy for perforated Crohn's disease up to 2 to3 months in the post operative period
  Groups: post operative Cronn's patients

SUMMARY:
crohn's disease patients who present by intestinal perforation as the first presentation are hard to deal with. Surgical techniques as anastmosis or diversion stoma and active course of the disease may greatly affect the quality of life. In post-operative period, is the priority to avoid the post operative complications and to improve surgical outcomes or to stop active course of the disease and to induce remission?. So, those patients were classified into two groups. one group received biological therapy early post operative and the other group received it 2 or 3 months later after surgery and the investigators will compare results between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* patients at or above 18 years old
* patients with perforated bowel diagnosed as Crohn's disease at presentation underwent surgery

Exclusion Criteria:

* patients less than 18 years old
* well known Crohn's disease patients on medical treatment
* associated bowel disease as malignancy and diverticulosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with Crohn's disease presented with bowel perforation
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2015-07-09 (Actual); Primary Completion 2025-07-09 (Actual); Study Completion 2025-07-09 (Actual)

PRIMARY OUTCOMES:
size of intra-abdominal fluids or collection | from the first post-operative day to 2 months postoperatively
  size of peritoneal fluids will be measured by surface area in centimeter square ( weight x height) using ultrasound
bowel function | from the first post-operative day to 2 months postoperatively
  bowel function will be assessed by hearing intestinal sound using Stethoscope
fecal fistula | from the first post-operative day to 2 months postoperatively
  if found, its amount will be calculated per day using calibrated colostomy bag
skin maceration | from the first post-operative day to 2 months postoperatively
  skin maceration surface area will be calculated by (weight x height) in centimeter square using a ruler
body weight | from the first post-operative day to 2 months postoperatively
  weight gain or weight loss will be measured in kg
age | 2 hours before surgery
  age in years will be recorded
sex | 2 hours before surgery
  sex of patients (male or female) will be recorded

CONTACTS AND LOCATIONS:
Locations (1):
- Zagazig University Hospitals, Zagazig, Egypt

IPD SHARING:
Plan to Share IPD: No
data will be available on demand by contacting the principle investigator